CLINICAL TRIAL: NCT02334488
Title: Prospective Multicenter Randomized Openlabel Study to Evaluate the Benefit on Renal Function at 12months Post-transplantation of Immunosuppressive Treatment With Withdrawal of Calcineurin Inhibitor at 3months and Combining Mycophenolate Sodium-Everolimus Versus Tacrolimus-Everolimus, in Patients With de Novo Kidney Transplant
Brief Title: Study Evaluating the Benefit of Two Immunosuppressive Strategies on Renal Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMéTé
Record Dates: First submitted 2014-11-03; First posted 2015-01-08 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus-Tacrolimus (Active Comparator): * Tacrolimus (Prograf®) started at 0,1 mg/kg/day since Day0, then adapted to C0 concentration (4-7 ng/ml),
  * Everolimus (Certican®) started within 24h after reperfusion, to be adapted to C0 concentration (3-8 ng/ml).
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Everolimus-Mycophenolate sodium (Experimental): * Everolimus (Certican®) started within 24h after reperfusion, to be adapted to C0 concentration (3-8 ng/ml),
  * Tacrolimus (Prograg®) started at 0,1 mg/kg/day from J0 then to be adapted to C0 concentration (4-7 ng/ml), then replacement by mycophenolate sodium (Myfortic®) at M3 (3 months visit) started at 1440 mg/day.
  Interventions: Drug: Everolimus; Drug: Mycophenolate sodium

INTERVENTIONS:
Drug: Everolimus — Active Comparator
  Other Names: Certican®
Drug: Tacrolimus — Active Comparator
  Other Names: Prograg®
  Arms: Everolimus-Tacrolimus
Drug: Mycophenolate sodium — Experimental Arm
  Other Names: Myfortic®
  Arms: Everolimus-Mycophenolate sodium

SUMMARY:
Prospective, multicenter, randomized and open label study evaluating the benefit on renal function at 12 months post-transplantation, with an immunosuppression without calcineurin inhibitor at 3 months and combining mycophenolate sodium-Everolimus versus an immunosuppression combining Everolimus-Tacrolimus, in de novo renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a first kidney transplant from a cadaveric or living donor

Exclusion Criteria:

* Double transplant
* Patient who has been treated with an immunosuppressive drug or study drug during the four weeks before administration of the first dose of Everolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Renal function as measured by estimated glomerular filtration rate GFR | One year after inclusion
  GFR unit : mL / min / 1.73 m2

CONTACTS AND LOCATIONS:
Overall Officials: Antoine THIERRY, MD, Principal Investigator — Poitiers University Hospital
Locations (14):
- France (14):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Caen University Hospital, Caen
  - Clermont Ferrand University Hospital, Clermont-Ferrand
  - Limoges University Hospital, Limoges
  - Georges Pompidou European Hospital, Paris
  - Necker Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Reims University Hospital, Reims
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Strasbourg University Hospital, Strasbourg
  - Tours University Hospital, Tours